CLINICAL TRIAL: NCT06040138
Title: Monitoring of Breathing Effort Through Pressure Time Product Measurement Using Airway Occlusion Pressure
Acronym: PTPPocc
Status: Recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: HOSPITAL BRITANICO DE BUENOS AIRES (Other); Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other); Sanatorio Anchorena San Martin (Other)
Responsible Party: Principal Investigator, EMILIO MARTIN STEINBERG, Principal Investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 6810
Record Dates: First submitted 2023-09-05; First posted 2023-09-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Failure; Weaning Failure
Keywords: mechanical ventilation; weaning; breathing effort; occlusion pressure; pressure time product; pressure support ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with prolonged weaning: Patients who have failed more than 3 spontaneous breathing trials, in pressure support ventilation, with hemodynamic and metabolic stability, and a regular and stable ventilatory pattern.
  Interventions: Diagnostic Test: End expiratory occlusion maneuver

INTERVENTIONS:
Diagnostic Test: End expiratory occlusion maneuver — An end expiratory occlusion maneuver will be performed during pressure support ventilation in patients with prolonged weaning.

SUMMARY:
Mechanical ventilation is essential in the management of patients in Intensive Care. The approach to patients with prolonged weaning is challenging.In this context, it is vital to implement "diaphragmatic protection" strategies, which consist of programming the level of ventilator assistance focused on sustaining the muscular effort within an objective range. The reference method for measuring inspiratory effort is the Pressure-Time Product (PTP) of the esophagus.

Recently, Bertoni et al. proposed the measurement of Occlusion Pressure as a non-invasive method, without the need to assess esophageal pressure, to estimate the magnitude of the effort and program assistance. Although it is a validated measurement for quantifying effort, it does not consider the duration of the effort performed by the patient, as well as the respiratory rate, two fundamental variables in terms of tolerance to the load. Therefore, the investigators propose the following study that will seek to validate the measurement of PTP in from the Occlusion Pressure, but considering inspiratory time and respiratory rate to obtain PTP per breath and per minute.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is an essential support in the management of patients in Intensive Care Units (ICU). According to international epidemiological studies, around 40% of patients admitted to ICU require ventilatory support.

International epidemiological data indicate that just over 55% of ICU patients are weaned from MV prematurely, and that approximately 20% experience difficult and prolonged weaning. In Argentina, our country, there are reports that this population amounts to 49.3%. One common denominator in the literature, international and national, regarding this section, is that such patients have more days of MV, ICU and hospital stay.

During prolonged weaning, monitoring of muscular effort becomes essential: both excessive and deficient efforts usually lead to diaphragmatic dysfunction. The former predisposes to fatigue, while the latter to atrophy. In this context, it is vital to implement "diaphragmatic protection" strategies, which consist of programming the level of assistance with a focus on muscular effort or muscular pressure (PMUS) to keep it within a target range.

The reference method for measuring inspiratory effort is the Pressure-Time Product of the esophagus (PTPESO), which involves the magnitude of PMUS measured through the change in esophageal pressure (PES) generated during inspiration, its duration, and respiratory rate (RR). For patients on partial ventilatory support, a PTP of 50 to 150 cmH2O/sec/min is recommended. Thus, PES becomes an everyday and reference tool for the management of patients with prolonged weaning from MV.

Recently, Bertoni et al. proposed measuring Occlusion Pressure (POCC) as a non-invasive method, i.e., without the need to evaluate PES, to estimate the magnitude of PMUS and program assistance in PSV. By means of a tele-expiratory occlusion maneuver of the airway, the maximum negative deflection of the signal during the patient's inspiration is quantified. This maneuver is called POCC. Then, through a simple multiplication by a constant, the value of PMUS in one cycle is obtained. Given the ease of measurement and its non-invasive nature, this technique has taken a leading role in the approach to patients during partial support at present.

Although the POCC is validated to quantify breathing effort, it has significant weaknesses. Some of these are that it only values the maximum deflection in an average of efforts, does not consider the time that the effort made by the patient lasts, nor the respiratory rate, two fundamental variables in terms of tolerance to the load (duration of contraction and frequency of repetition).

In this context, having a method that can estimate PTPESO non-invasively would be extremely useful to titrate the level of assistance in the framework of diaphragmatic protection strategies in patients with difficulties in being weaned from MV.

Therefore, the investigators propose the following study that will validate the measurement of PTPESO based on POCC, but considering the inspiratory time and respiratory rate to obtain PTP per breath and per minute. These variables will be called PTPPOCC-br and PTPPOCC-min, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mechanical ventilation, who failed 3 or more spontaneous breathing trials
* Esophageal balloon placed
* Who can trigger the ventilator
* With hemodynamic stability
* with P/F ratio above 150

Exclusion Criteria:

* under 18 years old of age
* pregnancy
* do not resuscitate order or expected poor short term prognosis
* refuse to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age with prolonged weaning from mechanical ventilation, who are in the intensive care units of the following hospitals: Hospital Italiano, Hospital Británico, Centro de Educación Médica e Investigaciones Clínicas 'Norberto Quirno' and Sanatorio Anchorena de San Martín, will be included
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Airway Occlusion Pressure | At the end of the study, estimated in July 2024
  An inspiratory pressure will be set to obtain a muscular pressure value of 8 to 12 cmH2O. This phase will be called PSV100%. After 15 minutes, the level of assistance will be modified by 50%, up or down, according to the result of the randomization, and vice versa, always considering the initial value. Each of these phases will be called PSV150% and PSV50% respectively, and will last 15 minutes. During the last 3 minutes, 3 end-expiratory occlusion at a rate of 1 maneuver per minute will be performed, in order to obtain the airway Occlusion Pressure.

SECONDARY OUTCOMES:
Esophageal Pressure Time product per breath (PTPESOF-br) and per minute (PTPESOF-min) | At the end of the study, estimated in July 2024
  Both the PTPESOF - br and the PTPESOF - min will be obtained directly from FluxReview, which calculates it automatically. To do this, the operator must select the desired breaths and load the value of the chest compliance (CCW) as input. For the correct estimation of this parameter, the value derived from the estimated vital capacity of the patient will be used, a method described by Mauri et al. and used in similar studies. [16] Segments of the PES signal in which erratic values or with artifacts are present will be excluded from the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Steinberg, RT, Principal Investigator — Hospital Italiano
Locations (4):
- Argentina (4):
  - Centro de Educación Médica e Investigaciones Clínicas "Norberto Quirno", Buenos Aires
  - Hospital Británico, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Sanatorio Anchorena San Martín, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Bertoni M, Telias I, Urner M, Long M, Del Sorbo L, Fan E, Sinderby C, Beck J, Liu L, Qiu H, Wong J, Slutsky AS, Ferguson ND, Brochard LJ, Goligher EC. A novel non-invasive method to detect excessively high respiratory effort and dynamic transpulmonary driving pressure during mechanical ventilation. Crit Care. 2019 Nov 6;23(1):346. doi: 10.1186/s13054-019-2617-0. PMID 31694692
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Brault C, Mancebo J, Suarez Montero JC, Bentall T, Burns KEA, Piraino T, Lellouche F, Bouchard PA, Charbonney E, Carteaux G, Maraffi T, Beduneau G, Mercat A, Skrobik Y, Zuo F, Lafreniere-Roula M, Thorpe K, Brochard L, Bosma KJ. The PROMIZING trial enrollment algorithm for early identification of patients ready for unassisted breathing. Crit Care. 2022 Jun 23;26(1):188. doi: 10.1186/s13054-022-04063-4. PMID 35739553
- [Background] Brochard L, Martin GS, Blanch L, Pelosi P, Belda FJ, Jubran A, Gattinoni L, Mancebo J, Ranieri VM, Richard JC, Gommers D, Vieillard-Baron A, Pesenti A, Jaber S, Stenqvist O, Vincent JL. Clinical review: Respiratory monitoring in the ICU - a consensus of 16. Crit Care. 2012 Dec 12;16(2):219. doi: 10.1186/cc11146. PMID 22546221
- [Background] Collett PW, Perry C, Engel LA. Pressure-time product, flow, and oxygen cost of resistive breathing in humans. J Appl Physiol (1985). 1985 Apr;58(4):1263-72. doi: 10.1152/jappl.1985.58.4.1263. PMID 3988680
- [Background] Combes A, Costa MA, Trouillet JL, Baudot J, Mokhtari M, Gibert C, Chastre J. Morbidity, mortality, and quality-of-life outcomes of patients requiring >or=14 days of mechanical ventilation. Crit Care Med. 2003 May;31(5):1373-81. doi: 10.1097/01.CCM.0000065188.87029.C3. PMID 12771605
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Dianti J, Fard S, Wong J, Chan TCY, Del Sorbo L, Fan E, Amato MBP, Granton J, Burry L, Reid WD, Zhang B, Ratano D, Keshavjee S, Slutsky AS, Brochard LJ, Ferguson ND, Goligher EC. Strategies for lung- and diaphragm-protective ventilation in acute hypoxemic respiratory failure: a physiological trial. Crit Care. 2022 Aug 29;26(1):259. doi: 10.1186/s13054-022-04123-9. PMID 36038890
- [Background] Dorado JH, Navarro E, Plotnikow GA, Gogniat E, Accoce M; EpVAr Study Group. Epidemiology of Weaning From Invasive Mechanical Ventilation in Subjects With COVID-19. Respir Care. 2023 Jan;68(1):101-109. doi: 10.4187/respcare.09925. Epub 2022 Nov 15. PMID 36379638
- [Background] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Background] Goligher EC, Dres M, Patel BK, Sahetya SK, Beitler JR, Telias I, Yoshida T, Vaporidi K, Grieco DL, Schepens T, Grasselli G, Spadaro S, Dianti J, Amato M, Bellani G, Demoule A, Fan E, Ferguson ND, Georgopoulos D, Guerin C, Khemani RG, Laghi F, Mercat A, Mojoli F, Ottenheijm CAC, Jaber S, Heunks L, Mancebo J, Mauri T, Pesenti A, Brochard L. Lung- and Diaphragm-Protective Ventilation. Am J Respir Crit Care Med. 2020 Oct 1;202(7):950-961. doi: 10.1164/rccm.202003-0655CP. PMID 32516052
- [Background] Jonkman AH, Rauseo M, Carteaux G, Telias I, Sklar MC, Heunks L, Brochard LJ. Proportional modes of ventilation: technology to assist physiology. Intensive Care Med. 2020 Dec;46(12):2301-2313. doi: 10.1007/s00134-020-06206-z. Epub 2020 Aug 11. PMID 32780167
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Mauri T, Yoshida T, Bellani G, Goligher EC, Carteaux G, Rittayamai N, Mojoli F, Chiumello D, Piquilloud L, Grasso S, Jubran A, Laghi F, Magder S, Pesenti A, Loring S, Gattinoni L, Talmor D, Blanch L, Amato M, Chen L, Brochard L, Mancebo J; PLeUral pressure working Group (PLUG-Acute Respiratory Failure section of the European Society of Intensive Care Medicine). Esophageal and transpulmonary pressure in the clinical setting: meaning, usefulness and perspectives. Intensive Care Med. 2016 Sep;42(9):1360-73. doi: 10.1007/s00134-016-4400-x. Epub 2016 Jun 22. PMID 27334266
- [Background] Penuelas O, Muriel A, Abraira V, Frutos-Vivar F, Mancebo J, Raymondos K, Du B, Thille AW, Rios F, Gonzalez M, Del-Sorbo L, Ferguson ND, Del Carmen Marin M, Pinheiro BV, Soares MA, Nin N, Maggiore SM, Bersten A, Amin P, Cakar N, Suh GY, Abroug F, Jibaja M, Matamis D, Zeggwagh AA, Sutherasan Y, Anzueto A, Esteban A. Inter-country variability over time in the mortality of mechanically ventilated patients. Intensive Care Med. 2020 Mar;46(3):444-453. doi: 10.1007/s00134-019-05867-9. Epub 2020 Jan 7. PMID 31912203
- [Background] Su PL, Kao PS, Lin WC, Su PF, Chen CW. Limited predictability of maximal muscular pressure using the difference between peak airway pressure and positive end-expiratory pressure during proportional assist ventilation (PAV). Crit Care. 2016 Nov 27;20(1):382. doi: 10.1186/s13054-016-1554-4. PMID 27888836